CLINICAL TRIAL: NCT01486654
Title: Transcranial Direct Current Stimulation and Aphasia Language Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Leora Cherney, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-kaye; 1R21DC009876-01A1 (NIH)
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Nonfluent Aphasia; Stroke
Keywords: Cortical stimulation; Ischemic Stroke; Aphasia; Speech and Language Rehabilitation
MeSH Terms: conditions — Aphasia, Broca; Stroke; Ischemic Stroke; Aphasia; Speech | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Anodal stimulation (Active Comparator)
  Interventions: Device: Transcranial Direct Current Stimulation - Anodal stimulation
- Cathodal stimulation (Active Comparator)
  Interventions: Device: Transcranial Direct Current Stimulation - Cathodal stimulation
- Sham stimulation (Placebo Comparator)
  Interventions: Device: Transcranial Direct Current Stimulation - Sham stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation - Cathodal stimulation — Cathodal transcranial direct stimulation (tDCS) to the left hemisphere, 1.0 mA for 13 minutes, is received five days a week, for six weeks, during the initial 13 minutes of 90 minutes of speech-language treatment.
  Other Names: Cortical stimulation; Transcranial direct current stimulation
  Arms: Cathodal stimulation
Device: Transcranial Direct Current Stimulation - Anodal stimulation — Anodal transcranial direct stimulation (tDCS) to the left hemisphere, 1.0 mA for 13 minutes, is received five days a week, for six weeks, during the initial 13 minutes of 90 minutes of speech-language treatment.
  Other Names: Cortical stimulation; Transcranial direct current stimulation
  Arms: Anodal stimulation
Device: Transcranial Direct Current Stimulation - Sham stimulation — Sham stimulation provided together with 90 minutes of speech language therapy, 5 days a week, for 6 weeks.
  Other Names: No stimulation
  Arms: Sham stimulation

SUMMARY:
The purpose of this study is to evaluate the effectiveness of small amounts of electrical current, applied without surgery to the brain, in combination with speech-language treatment, on the language outcome of study subjects with nonfluent aphasia (i.e. difficulty with the comprehension and expression of spoken and written language) following a stroke.

DETAILED DESCRIPTION:
Stroke is the third leading cause of death and the most common cause of disability in the United States. According to the American Stroke Association, the prevalence of stroke in the U.S. is approximately 4.8 million with approximately 700,000 additional strokes occurring annually. Approximately 150,000 to 250,000 stroke survivors becoming severely and permanently disabled each year.

A common neurological deficit among stroke survivors, and thus a substantial contributor to post-stroke disability, is aphasia. The loss of, or difficulty with language is extremely debilitating and has enormous social and economic impact on quality of life. Presently, the only treatment available for persons with aphasia is speech-language rehabilitation.

With rehabilitation only, however, many patients achieve a less than satisfactory improvement in speech-language function, and thus are left with significant disability.

Enhancing stroke recovery by facilitating brain plasticity with the direct application of stimulation to the cerebral cortex is a new area of investigation and shows promise for improving language recovery in stroke-induced aphasia, most probably when it is combined with intense learning. There are several methods of delivering cortical brain stimulation to modulate cortical excitability, each of which have been studied in animal models with promising results, and subsequently applied to the rehabilitation of motor deficits after stroke. Applications to language problems after stroke are only emerging. Nevertheless, results suggest a potential role for cortical stimulation as an adjuvant strategy in aphasia rehabilitation.

Of the cortical stimulation methods available, transcranial direct current stimulation (tDCS) has the greatest potential for clinical use in view of its non-invasive application, ease of administration and relatively low cost. tDCS is a method of delivering weak polarizing electrical currents to the cortex via two electrodes placed on the scalp. The nature of the effect depends on the polarity of the current. Anodal tDCS has an excitatory effect; cathodal tDCS induces inhibition.

This study proposes to evaluate the safety, feasibility, and effectiveness of anodal and cathodal tDCS in study subjects with Broca's aphasia after stroke, delivered concurrent with speech-language rehabilitation.

Subjects will receive speech and language therapy combined with either anodal, cathodal, or sham stimulation applied to the lesioned left hemisphere. The polarity conditions will be compared with each other and with sham stimulation, to determine safety, the degree to which improvements in language performance occur, and the degree to which they are maintained over time.

The protocol is single-blind. Neither the subjects nor the outcomes assessor will know what stimulation the subject received until the study's conclusion; the investigator applying the stimulation will know.

ELIGIBILITY:
Inclusion Criteria:

* A single unilateral left-hemisphere infarct that is confirmed by CT scan or MRI
* Nonfluent aphasia, with a mean length of utterance of 0-4 words and an Aphasia Quotient score on the Western Aphasia Battery of 25-70
* Age 21 or older
* At least 6 months post-stroke
* Premorbidly right-handed, as determined by the Edinburgh Handedness Inventory
* Premorbidly literate in English
* Completed at least an eighth grade education
* Visual acuity no worse than 20/100 corrected in the better eye
* Auditory acuity, aided in the better ear, no worse than 30 dB HL on a pure tone hearing screening (conducted at 500, 1000, 2000, and 4000 Hz.)

Exclusion Criteria:

* Any other neurological condition (other than cerebral vascular disease) that could potentially affect cognition or speech, such as Parkinson's Disease, Alzheimer's Dementia, traumatic brain injury
* Any significant psychiatric history prior to the stroke, such as severe major depression or psychotic disorder requiring hospitalization; subjects with mood disorders who are currently stable on treatment will be considered
* Active substance abuse
* Seizure disorder that precludes safe participation in this trial
* Absence of left hemisphere activation during two of the three fMRI tasks
* Presence of lesions that encompass premotor cortex from the Sylvian fissure to a point high on the convexity

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Aphasia Quotient (AQ) on the Western Aphasia Battery | Change from Baseline in Western Aphasia Battery at 6 weeks

SECONDARY OUTCOMES:
Functional communication skills | Change from Baseline in functional communication skills at 6 weeks
  Scores derived from language sample analyses
Participation in everyday activities | Change from Baseline in participation in everyday activities at 6 weeks
  Measures on CETI, BOSS, CCRSA
Western Aphasia Battery - Reading and Writing scores | Change from Baseline in Western Aphasia Battery Reading and Writing scores at 6 weeks
Western Aphasia Battery Aphasia Quotient (Maintenance) | Change in Western Aphasia Battery AQ from 6 weeks to 12 weeks
Western Aphasia Battery Reading and Writing Scores (Maintenance) | Change in WAB Reading and Writing Skills from 6 weeks to 12 weeks
Functional Communication Skills (Maintenance) | Communication skills from 6 weeks to 12 weeks
Participation in everyday activities (Maintenance) | Change in participation in everyday activities from 6 weeks to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Leora R Cherney, PhD, Principal Investigator — Rehabilitation Institute of Chicago, Chicago, IL
Locations (1):
- Center for Aphasia Research & Treatment, Rehabilitation Institute of Chicago, Chicago, Illinois, United States